CLINICAL TRIAL: NCT05712668
Title: A Randomized, Controlled Trial for Asynchronous Telemedicine Use in Preoperative Counseling for Individuals With Endometrial Cancer
Brief Title: Telemedicine Use in Preoperative Counseling for Endometrial Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Shannon Armbruster, Assistant Professor, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 21-1305
Record Dates: First submitted 2023-01-02; First posted 2023-02-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Telemedicine; Counseling
Keywords: Telemedicine; Preoperative Counseling

STUDY DESIGN:
Intervention Model Description: A total of 100 patients will be enrolled and randomized if they meet the inclusion criteria. Fifty patients allocated will be allocated to receive pre-operative counseling via standard face-to-face care and 50 patients allocated to receive standard pre-operative counseling with the addition of asynchronous telemedicine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Pre-operative Counseling (Active Comparator): Participants will receive standard counseling.
  Interventions: Behavioral: Preoperative counseling
- Standard Pre-operative Counseling plus Asynchronous Telemedicine (Experimental): Participants will receive standard counseling plus access to a 5 minute video reviewing their in-office counseling.
  Interventions: Behavioral: Preoperative counseling; Behavioral: Asynchronous telemedicine

INTERVENTIONS:
Behavioral: Preoperative counseling — Providers will review the diagnosis, surgical planning, risks/benefits/alternatives to surgery, post-operative care, and long term scope of care.
Behavioral: Asynchronous telemedicine — An asynchronous video will be delivered by Mytonomy. This platform allows investigators to track user analytics relating to the time, frequency, or duration watched by the user.
  Other Names: Mytonomy
  Arms: Standard Pre-operative Counseling plus Asynchronous Telemedicine

SUMMARY:
To determine whether telemedicine is an acceptable addition to pre-operative counseling, compared to face-to-face communication alone for patients with endometrial cancer.

DETAILED DESCRIPTION:
Newly diagnosed endometrial cancer survivors, who are presenting for their initial consultation with a plan for minimally invasive surgery, will be randomized 1:1 to standard counseling or standard counseling plus asynchronous telemedicine video. The asynchronous video will be available outside of the office and can be viewed multiple times. The primary endpoint is patient anxiety, measured via the State-Trait Anxiety Inventory (STAI) questionnaire, assessed before surgery. The secondary outcomes of anxiety following surgery as well as patient satisfaction with counseling type (measured via the Patient Satisfaction Questionnaire (PSQ-18)) before and after surgery will be compared between groups. Both groups will complete questionnaires following their initial consultation (but before surgery) and at their post-operative visit. For the telemedicine group, the duration and frequency of video views will be collected. Participants completing both surveys will receive a survivorship gift bag.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical stage I histologically confirmed endometrial carcinoma, which is clinically confined to the uterus and comprises approximately two-thirds of all endometrial carcinoma cases
2. Patients undergoing planned minimally invasive surgical procedures, such as a minimally invasive technique such as conventional laparoscopy or robotic-assisted laparoscopy, as part of treatment at the Division of Gynecologic Oncology at Carilion Clinic, Roanoke, VA
3. Internet/cellular access at home
4. Ability to read and comprehend materials on questionnaires

Exclusion Criteria:

1 Patients that do not meet the inclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants have been diagnosed with endometrial cancer
Enrollment: 100 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety related to preoperative counseling | Following the initial office visit or online viewing session, prior to surgery
  It will be measured via the State-Trait Anxiety Inventory (STAI) questionnaire, a validated tool used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. STAI is comprised of 20 concise questions on a 4-point Likert scale.

SECONDARY OUTCOMES:
Patient satisfaction with preoperative counseling | Following the initial office visit or online viewing session, prior to surgery
  It will be measured via the Patient Satisfaction Questionnaire (PSQ-18), which is also a validated questionnaire. It is comprised of 18 questions, also on a Likert scale, used to assess 7 dimensions of patient satisfaction.
Patient satisfaction with preoperative counseling, surgical impact | At the postoperative exam, approximately 2-4 weeks from surgery
  It will be measured via the Patient Satisfaction Questionnaire (PSQ-18), which is also a validated questionnaire. It is comprised of 18 questions, also on a Likert scale, used to assess 7 dimensions of patient satisfaction.
Anxiety related to preoperative counseling, surgical impact | At the postoperative exam, approximately 2-4 weeks from surgery
  It will be measured via the State-Trait Anxiety Inventory (STAI) questionnaire, a validated tool used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes. STAI is comprised of 20 concise questions on a 4-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Armbruster, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States